CLINICAL TRIAL: NCT06176261
Title: DATO-BASE: A Phase 2 Trial of DATOpotamab-deruxtecan for Breast Cancer Brain metAstaSEs
Brief Title: DATO-BASE: DATOpotamab-deruxtecan for Breast Cancer Brain metAstaSEs
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sarah Sammons, MD (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor-Investigator, Sarah Sammons, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-533
Record Dates: First submitted 2023-12-07; First posted 2023-12-19 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Breast Cancer Female; Metastatic Triple-Negative Breast Carcinoma; ER Positive Breast Cancer; HER2-negative Breast Cancer; HER2 Negative Breast Carcinoma; ER-negative Breast Cancer
Keywords: Breast Cancer; Breast Cancer Female; Metastatic Triple-Negative Breast Carcinoma; ER Positive Breast Cancer; HER2 Negative Breast Cancer; HER2 Negative Breast Carcinoma; ER Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A: Estrogen Receptor Positive HER2-Negative Metastatic Breast Cancer (Experimental): 24 participants will be enrolled and will complete study procedures as outlined below:
  * Baseline visit with optional CSF collection via lumbar puncture and assessments.
  * CT or MRI scans every 6 weeks for 24 weeks, then every 9 weeks.
  * Cycle 1 Through End of Treatment:
    --Day 1 of 21 day cycle: Predetermined dose of Datopotamab Deruxtecan 1x daily.
  * End of Treatment:
    * Follow up every 6 months.
    * Optional CSF collection via lumbar puncture.
    * CT or MRI scans every 12 weeks.
  Interventions: Drug: Datopotamab Deruxtecan
- Cohort B: Metastatic Triple-Negative Breast Cancer (Experimental): 24 participants will be enrolled and will complete study procedures as outlined below:
  * Baseline visit with optional CSF collection via lumbar puncture and assessments.
  * CT or MRI scans every 6 weeks for 24 weeks, then every 9 weeks.
  * Cycle 1 Through End of Treatment:
    --Day 1 of 21 day cycle: Predetermined dose of Datopotamab Deruxtecan 1x daily.
  * End of Treatment:
    * Follow up every 6 months.
    * Optional CSF collection via lumbar puncture.
    * CT or MRI scans every 12 weeks.
  Interventions: Drug: Datopotamab Deruxtecan
- Cohort C: HER2-Negative Metastatic Breast Cancer (any ER Expression) with Leptomeningeal Metastases (Experimental): * Baseline visit with CSF collection via lumbar puncture and assessments.
  * CT or MRI scans every 6 weeks for 24 weeks, then every 9 weeks.
  * Cycle 1
    --Day 1 of 21 day cycle: Predetermined dose of Datopotamab Deruxtecan 1x daily.
  * Cycle 2
    * Day 1 of 21 day cycle: Predetermined dose of Dato-DXd 1x daily.
    * Day 2 of 21 day cycle: CSF collection.
  * Cycle 3 Through End of Treatment:
    --Day 1 of 21 day cycle: Predetermined dose of Datopotamab Deruxtecan 1x daily.
  * End of Treatment:
    * Follow up every 6 months.
    * Optional CSF collection via lumbar puncture.
    * CT or MRI scans every 12 weeks.
  Interventions: Drug: Datopotamab Deruxtecan

INTERVENTIONS:
Drug: Datopotamab Deruxtecan — Antibody-drug conjugate, 100 mg single-use vial, via intravenous infusion per protocol.
  Other Names: DS-1062; DS-1062a, Dato-DXd

SUMMARY:
The purpose of this study is to test the safety and effectiveness of the study drug datopotamab deruxtecan in participants with metastatic breast cancer that has spread to the brain.

The name of the study drug used in this research study is:

Datopotamab deruxtecan (a type of antibody-drug conjugate)

DETAILED DESCRIPTION:
This is a single-arm, multi-cohort, open-label, phase II trial designed to evaluate the safety and efficacy of datopotamab deruxtecan for the treatment of CNS metastases in patients with HER2-negative metastatic breast cancer.

Participants will be enrolled in three different groups: Cohort A for estrogen receptor (ER)-positive HER2-negative breast cancer, Cohort B for metastatic triple negative breast cancer, and Cohort C for HER2-negative metastatic breast cancer which has spread to the leptomeninges (which surround the brain or spinal cord).

Datopotamab deruxtecan is a new type of anti-cancer drug called an "antibody drug conjugate" (ADC) that targets cancer cells expressing a specific molecule on the tumor cell membrane.

The U.S. Food and Drug Administration (FDA) has not approved datopotamab deruxtecan as a treatment for metastatic, Human epidermal growth factor receptor-2 (HER2) negative breast cancer.

The research study procedures include screening for eligibility, blood tests, questionnaires, and study treatment visits, Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) scans, electrocardiograms, echocardiograms, and cerebral spinal fluid (CSF) collection.

It is expected that about 58 people will take part in this research study.

Daiichi Sankyo Inc. is funding this study and providing the study drug, datopotamab deruxtecan.

ELIGIBILITY:
Inclusion Criteria :

* Metastatic breast cancer that is pathologically confirmed to be HER2-negative according to 2018 ASCO/CAP guidelines 55.
* Radiological confirmation of metastatic disease.
* Cohorts A and B: Presence of newly diagnosed brain metastases or brain metastases progressing after prior local and/or systemic therapy.
* Cohorts A and B: Participants must have a baseline MRI of the brain performed with and without gadolinium contrast, and must have central nervous system metastases with at least one measurable brain metastasis ≥ 1.0 cm in size (per RANO-BM) that has not been irradiated, or has progressed despite prior radiation therapy and/or systemic therapy (in the opinion of the treating physician). For cohorts A and B, head CT with contrast may be used in place of MRI at baseline and throughout the trial if MRI is contraindicated and the participant's CNS metastases are clearly measurable by head CT.
* Cohorts C: Radiological evidence of evaluable leptomeningeal disease and clinical diagnosis of LMD per treating investigator. A positive CSF cytology is not required.
* Cohort A: prior progression to treatment with at least one line of endocrine treatment (with or without CDK4/6 inhibition) in the metastatic setting is mandatory. Patients experiencing recurrence during adjuvant endocrine treatment will be also considered eligible for the trial. There is no limit on the number of prior lines acceptable for the purpose of enrollment in this study.
* Cohort B and C: no prior treatment is required (i.e., previously untreated patients are eligible). There is no limit on the number of prior lines of therapy acceptable for the purpose of enrollment in this study.
* Participants may have measurable or non-measurable extracranial disease. Participants are NOT required to have extracranial disease, but must have imaging done to document disease status at baseline.
* Age ≥ 18 years.
* ECOG Performance Status 0-2
* Participants must have adequate treatment washout period before registration, defined as > 4 weeks from major surgery, > 2 weeks from radiation treatment. For weekly chemotherapy regimens, > 2 weeks from chemotherapy; for every 3 weekly regimens, > 3 weeks from chemotherapy. At least 2 weeks from other systemic or targeted or investigational therapies (other than endocrine therapy) for breast cancer. No washout is required for endocrine therapy (e.g. aromatase inhibitors, tamoxifen, fulvestrant) but patients should discontinue prior to start of protocol therapy. Patients on ovarian suppression are allowed (but not required) to continue ovarian suppression at the discretion of their treating provider.
* Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
* Adequate organ function as defined by the following values:

  * Hemoglobin ≥ 9.0 g/dL. Red blood cell/plasma transfusion is not permitted within 1 week prior to screening assessment.
  * Absolute neutrophil count ≥1,500/mm3. Granulocyte colony-stimulating factor administration is not permitted within 1 week prior to screening assessment.
  * Platelets ≥100,000/mm3. Platelet transfusion is not permitted within 1 week prior to screening assessment.
  * Total bilirubin ≤ 1.5 institutional ULN if no liver metastases; or ≤ 3 x ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline.
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN OR ≤ 5.0 x institutional ULN for patients with documented liver metastases
  * Serum creatinine ≤ 1.5 mg/dL (or glomerular filtration rate ≥ 30 ml/min as determined by the Cockcroft-Gault equation)
* Participants with a history of chronic viral conditions such as HIV, Hepatitis B/C, should not be systemically excluded but have thoughtful consideration of inclusion, unless safety is a concern. Testing for these conditions is not required at baseline.
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 14 days of initiating protocol therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Visceral crisis or impending visceral crisis
* CNS complications for whom urgent neurosurgical intervention is indicated (i.e., resection, shunt placement)
* Indication for immediate local therapy to CNS lesion(s) as defined by local standard
* Evidence of significant (i.e., symptomatic) intracranial hemorrhage

  -> 2 seizures within 4 weeks prior to study entry (registration)
* Ongoing/persistent toxicities caused by previous anti-cancer therapy (except alopecia) not yet improved to Grade ≤ 1 OR baseline prior to study entry (registration)
* Known contraindication to MRI (e.g., due to pacemaker, ferromagnetic implants, claustrophobia, extreme obesity, hypersensitivity). However, for cohorts A and B, head CT with contrast may be used in place of MRI at baseline and throughout the trial if MRI is contraindicated and the participant's CNS metastases are clearly measurable by head CT.
* Concurrent administration of other anti-cancer therapy during the course of this study is not allowed. Concurrent use of supportive care medications is allowed, and certain medications are required (see Section 5.1).
* Uncontrolled intercurrent illness, including (but not limited to) active infection, severely compromised pulmonary function, unstable angina pectoris, uncontrolled cardiac arrhythmia, active ischemic heart disease, myocardial infarction within the previous six months, gastric or duodenal ulceration diagnosed within the previous six months, chronic liver or renal disease, or severe malnutrition. Note that if a patient has controlled diabetes mellitus, but is unable to monitor blood glucose at home, they will be excluded from the trial.
* Participants must not have a condition requiring ongoing systemic treatment with corticosteroids (>4 mg daily dexamethasone (or bioequivalent)) or other immunosuppressive medications within 7 days prior to the baseline MRI. Corticosteroids administration must be stable and planned to remain ≤ 4 mg daily for the duration of protocol treatment. However, use of corticosteroids for clinical symptoms is allowed based upon treating physician discretion.
* History of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
* A history of uncontrolled seizures, CNS disorders, or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs.
* A history of malignancy other than breast cancer, except (a) adequately resected non-melanoma skin cancer, (b) curatively treated in situ disease, or (c) other solid tumors curatively treated, with no evidence of disease for ≥ 3 years.
* Major surgery, open biopsy, or significant traumatic injury within 28 days prior to the initiation of protocol therapy, or anticipation of need for a major surgical procedure during the study.
* Clinically significant corneal disease.
* Has a history of severe hypersensitivity reactions to either the drug or inactive ingredients (including but not limited to polysorbate 80) of datopotamab deruxtecan.
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Negative pregnancy test (urine and/or serum) is required for women of childbearing potential. Pregnant or lactating women are excluded from participation due to potential teratogenic effects of study drug.
* Female participants must be either:

  * post-menopausal for at least 1 year
  * surgically sterile, or
  * if of childbearing potential and sexually active with a non-sterilized male partner, must agree to use one highly effective form of birth control for the entire treatment period and for at least 7 months after the last dose of datopotamab deruxtecan (see Section 5.4 for complete list of highly effective birth control methods).
* Female participants must not donate, or retrieve for their own use, ova at any time during this study and for at least 7 months after the last dose of datopotamab deruxtecan.
* Female participants must refrain from breastfeeding while on study and for at least 7 months after the last dose of datopotamab deruxtecan.
* Male participants who intend to be sexually active with a female partner of childbearing potential must be surgically sterile or using an acceptable method of contraception (see Section 5.4 for complete list of highly effective birth control methods) from the time of screening throughout the total duration of the study and the drug washout period (at least 4 months after the last dose of study intervention) to prevent pregnancy in a partner. Male participants must not donate or bank sperm during this same time period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) in RANO-BM Criteria | 3 years
  The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RANO-BM criteria defined protocol section 11.1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 3 years
  The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECISTv1.1 criteria.
Clinical Benefit Rate at 18 weeks (CBR18) | 18 Weeks
  CBR defined as proportion of participants with defined as intracranial CR, intracranial PR, or stable disease (SD) in both intracranial and extracranial sites ≥ 18 (CBR18) . In the case of intracranial CR or PR, to be considered clinical benefit, extracranial disease must also be stable or better at the time of intracranial response. CBR will be reported for Cohort A and Cohort B only
Clinical Benefit Rate at 24 weeks (CBR24) | 24 Weeks
  CBR defined as proportion of participants with defined as intracranial CR, intracranial PR, or stable disease (SD) in both intracranial and extracranial sites ≥ 24 (CBR24) . In the case of intracranial CR or PR, to be considered clinical benefit, extracranial disease must also be stable or better at the time of intracranial response. CBR will be reported for Cohort A and Cohort B only
Median Progression-Free Survival (PFS) | Assessed from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, up to 3 years
  Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) defined per RANO-BM criteria. or death, or is censored at time of last disease assessment.
Median Overall Survival (OS) | Assessed from date of enrollment until the date of death from any cause, up to 3 years
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Site of First Progression | Assessed from date of enrollment until the date of first progression from any cause, up to 3 years
  Site of first progression defined as the number of participants has progression in each sites. Progression defined per RANO-BM criteria.
Grade 3-5 Treatment-related Toxicity Rate | From time of first dose of study treatment through 30 days after last dose of treatment, up to 3 years
  All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 that are not resolved in accordance with treatment guidelines were counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Sammons, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Miami Baptist Cancer Institute/, Miami, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
URL: https://www.dana-farber.org/research/innovations